CLINICAL TRIAL: NCT02566499
Title: Performance Assessment of a First Generation Breast Microwave Imaging System: Study of Breast Abnormalities Detection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Improved algorithms have resulted in a proposed redesign of detection system. Once completed, a new trial will be planned.
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B2015:73
Record Dates: First submitted 2015-07-13; First posted 2015-10-02 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Breast Diseases
Keywords: Medical imaging; Microwaves
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abnormal x-ray Mammography group (Experimental): A Breast Microwave Imaging Procedure will be carried out on volunteers who have abnormal x-ray mammograms, prior to the volunteer undergoing a biopsy to confirm diagnosis (as part of their normal care).
  Interventions: Device: Breast Microwave Imaging

INTERVENTIONS:
Device: Breast Microwave Imaging — A Breast Microwave Imaging Procedure will be carried out on volunteers who have abnormal x-ray mammograms, prior to the volunteer undergoing a biopsy to confirm diagnosis (as part of their normal care).

SUMMARY:
The main goal of this project is to assess the ability of a recently developed Breast Microwave Imaging (BMI) system to detect abnormalities in a human breast. These trials will be performed by recruiting fourteen volunteers that have been diagnosed with breast abnormalities using x-ray mammography. The breast presenting the abnormality will be imaged using the BMI system in a controlled and comfortable environment. As this is a feasibility study of the technology, and has the main goal to evaluate the diagnostic accuracy of this technology. The data collected from this study will be used to: (1) evaluate the overall participant experience during the BMI imaging procedure, (2) optimize the design of the BMI imaging system (both hardware and software), (3) open discussions with other medical professionals (e.g. radiologists) about the clinical feasibility of this emerging diagnostic imaging modality.

DETAILED DESCRIPTION:
The Breast Microwave Imaging (BMI) system that will be used in this study is designed to detect breast abnormalities using low power microwave waveforms. The system is formed by three main components:

1. Patient bed. The volunteer will be positioned in this bed in a prone position where with the breast to be imaged in a pendant position.
2. Instrumentation rack. This component contains all the microwave instrumentation and motion mechanisms required to illuminate the breast using an ultrawide band waveform and record the responses from the breast structures.
3. Control computer. This component is used to control the motion of the mechanical components of the system and to retrieve the responses from the breast structures from the microwave instruments and store them in an electronic format.

The system takes between 7.5 to 10 minutes to collect a three dimensional dataset from a single breast.

The BMI system used in the study operates in the frequency range of 20 megahertz (MHz) to 9 gigahertz (GHz). Canadian safety limits for the interaction of these non-ionizing electromagnetic waves with humans are outlined in the Health Canada publication "Safety Code 6: Limits of Human Exposure to Radiofrequency Electromagnetic Energy in the Frequency Range from 3 kilohertz (kHz) to 300 GHz [1]. For unregulated environments, the Specific Absorption Rate (SAR) limit set by Health Canada is 1.6 W/Kg. In the system used in this study, radio-frequency energy is generated via the Vector Network Analyzer (VNA). If the VNA is set at its maximum output power, which is 3.2 milliwatt (mW), the power received at 5 cm from the antenna (which is the distance where the breast will be) was measured to be 890 microwatt, which would yield a SAR value of 0.0196 W/kg.

References

[1] Consumer and Clinical Radiation Protection Bureau, Limits of Human Exposure to Radiofrequency Electromagnetic Energy in the Frequency Range from 3 kHz to 300 GHz, Health Canada, Ottawa, Ontario, 2015.

ELIGIBILITY:
Inclusion Criteria:

* The volunteers must be at least 40 years old.
* The volunteers should have been diagnosed with a breast abnormality using x-ray mammography within the preceding two months.

Exclusion Criteria:

* The volunteers should not have breast implants.
* The volunteers should have not yet had a biopsy.

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy (NO units) | 1 year
  Diagnostic Accuracy = (TP+TN)/(TP+FP+FN+TN): The fraction of patients that are diagnosed accurately, which is in turn a function of the Sensitivity and Specificity of the test.
  Sensitivity: The probability that a test result will be positive when the disease is present (true-positive fraction) = TP/(TP+FN)
  Specificity: The probability that a test result will be normal when the disease is absent (true-negative fraction) = TN/(FP+TN)
  TP = True Positive TN = True Negative FP = False Positive FN = False Negative

SECONDARY OUTCOMES:
Sensitivity (NO units) | 1 year
  Sensitivity: The probability that a test result will be positive when the disease is present (true-positive fraction) = TP/(TP+FN)
  TP = True Positive TN = True Negative FP = False Positive FN = False Negative
Specificity (NO units) | 1 year
  Specificity: The probability that a test result will be normal when the disease is absent (true-negative fraction) = TN/(FP+TN)
  TP = True Positive TN = True Negative FP = False Positive FN = False Negative

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pistorius, Ph.D., Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: No